CLINICAL TRIAL: NCT06122584
Title: Prospective, Multi-Center Study to Assess the Diagnostic Performance of [18F]PSMA-1007 PET/CT Imaging in Patients With Newly-Diagnosed High-Risk or Very-High-Risk Prostate Cancer
Brief Title: Diagnostic Performance of [18F]PSMA-1007 PET/CT Imaging in Patients With Newly-Diagnosed Prostate Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ABX advanced biochemical compounds GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EAGLE-i
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]PSMA-1007 (Experimental): Single intravenous administration of [18F]PSMA-1007 for Positron Emission Tomography (PET) scan
  Interventions: Drug: [18F]PSMA-1007

INTERVENTIONS:
Drug: [18F]PSMA-1007 — Diagnostic radiopharmaceutical for PET scan

SUMMARY:
This study assess the Diagnostic Performance of [18F]PSMA-1007 PET/CT Imaging in Patients with Newly-Diagnosed High-Risk or Very-High-Risk Prostate Cancer

ELIGIBILITY:
Inclusion Criteria:

1. The patient (male) is aged 18 years or above.
2. The patient is able to understand the information presented to him concerning the nature, scope, and consequences of the trial as set out in the information provided to the patient AND has provided written informed consent to participate.
3. The patient has newly diagnosed, biopsy-proven, clinically localized prostate adenocarcinoma, and curative prostatectomy with extended pelvic lymph node dissection is his preferred course of treatment.
4. The patient has at least high-risk disease as defined by the NCCN guidelines (version 1.2023). That is, the presence of any one or more of the following:

   * Overall ISUP grade group 4 or 5,
   * Clinical category T3a or greater,
   * Serum PSA level greater than 20 ng/ml.
5. The patient has undergone conventional imaging (CT or MRI, and bone scan if clinically indicated) to detect the presence of pelvic nodal involvement and bone or visceral metastases within 60 days of the planned PET-CT procedure.

Exclusion Criteria:

1. Patients for whom radical prostatectomy is not clinically appropriate or the patient is otherwise unlikely to undergo radical prostatectomy with extensive pelvic lymph node dissection.
2. The patient has received any therapy - be it radiation, surgical or drug therapy - for his prostate cancer.
3. The patient has any contraindication(s) for and/or known hypersensitivity to any constituent(s) of [18F]PSMA-1007.
4. The patient is not able to have PET-CT scans (for example, because of weight, claustrophobia, or inability to lie still for the duration of the scan).
5. The patient is closely affiliated to the investigation site; e.g. is a first-degree relative of the investigator.
6. At the time of screening, the patient is receiving any other investigational agent(s), or he has received any such agent(s) within the previous 30 days, or he is scheduled to receive any such agent(s) in the period up to the planned date for the last study visit.
7. The patient has previously been enrolled in this trial.
8. The patient has previously undergone PET imaging with any PSMA-avid product.
9. The patient has histological evidence of small-cell carcinoma of the prostate.
10. The patient is clinically unstable or requires emergency treatment.
11. The patient has any mental condition rendering him incapable of understanding the nature, scope, and consequences of the trial as set out in the information given to the patient.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of [18F]PSMA-1007 PET/CT for the detection of pelvic nodal disease (N1) compared to histology as the standard of reference | 6 to 8 weeks post-surgery

CONTACTS AND LOCATIONS:
Locations (18):
- CHRU de Nancy, Nancy, France
- Germany (8):
  - Carl Gustav Carus Faculty of Medicine, TUD Dresden, Dresden
  - University Hospital Düsseldorf, Düsseldorf
  - St. Antonius Hospital, Gronau
  - University Hospital Hamburg-Eppendorf, Hamburg
  - University Hospital Leipzig, Leipzig
  - Klinikum rechts der Isar, TUM, München
  - University Hospital Münster, Münster
  - Universitätsmedizin Rostock, Rostock
- Italy (2):
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori", Meldola
  - IRCCS Ospedale Sacro Cuore-Don Calabria, Verona
- Japan (2):
  - The University of Osaka Hospital, Osaka
  - National Cancer Center, Tokyo
- Netherlands (2):
  - CWZ, Nijmegen
  - Radboud UMC, Nijmegen
- Spain (3):
  - Hospital Del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Vithas Valencia 9 de Octubre, Valencia